CLINICAL TRIAL: NCT06517082
Title: An EHR-embedded Pragmatic Stepped-wedge Individual Randomized Clinical Trial of Ambient Artificial Intelligence to Improve Provider Well-Being
Brief Title: Ambient AI for Provider Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-1028; A534285 (Other: UW- Madison); Protocol Version 7/7/2024 (Other: UW- Madison)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthcare Provider Well-being
Keywords: Artificial Intelligence; Physician well-being; Healthcare provider
MeSH Terms: interventions — Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: The stepped wedge design involves staggered implementation of an intervention across different providers over multiple time periods, allowing all providers to eventually receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ambient Listening Group 1 (Experimental): Participants randomized to this arm will start using Ambient AI at week 7.
  Interventions: Other: Artificial Intelligence
- Ambient Listening Group 2 (Experimental): Participants randomized to this arm will start using Ambient AI at week 13.
  Interventions: Other: Artificial Intelligence
- Ambient Listening Group 3 (Experimental): Participants randomized to this arm will start using Ambient AI at week 19.
  Interventions: Other: Artificial Intelligence

INTERVENTIONS:
Other: Artificial Intelligence — Ambient AI software intervention is implemented into the providers workflow. The software incorporates Automated Speech Recognition technology with Large Language Models to generate clinical documentation in real-time.

SUMMARY:
The goal of this clinical trial is to learn whether using Ambient Artificial Intelligence for provider documentation will enhance provider well-being and improve documentation quality.

Participants will complete their documentation using the Ambient AI software.

DETAILED DESCRIPTION:
Provider documentation of patient visits is a time-consuming activity that extends throughout the workday and often continues outside office hours. This ongoing clerical burden negatively impacts provider well-being, contributing to burnout and job dissatisfaction.

To address these challenges, the researchers propose to test the effectiveness of the Ambient AI tool in improving provider fulfillment and note documentation efficiency. The overarching goal is to leverage AI technology to enhance provider well-being and documentation quality.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare Provider in the UW Health Outpatient Clinic Setting
* Willingness to engage and use ambient technology
* Owns an Apple mobile device, as the software is accessible only on this platform
* Adult (greater than 18 years)
* English or Spanish speaking
* Completed the training and in-servicing required to use the tool
* Providing outpatient care to no less than 20 encounters on a weekly average

Exclusion Criteria:

* Planned leave in 6 weeks following randomization
* Not registered onto Epic's mobile Haiku system for access
* Enrolled in a virtual scribe program and not willing to leave the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Change in provider fulfillment index | Baseline to weeks 6, 12, 18, and 24
  Using the Professional Well-Being Academic Consortium Survey Measures, the fulfillment index is a 6-item questionnaire. Each question is scored on a 0-4 Likert scale, with total possible scores of 0-24. Higher scores indicate greater fulfillment
Change in provider burnout | Baseline to weeks 6, 12, 18, and 24
  Using the Professional Well-Being Academic Consortium Survey Measures, the burnout index includes two subcomponents of work exhaustion and interpersonal disengagement. It is a 10-item questionnaire, scored together as a composite. Each question is scored on a 0-4 Likert scale, with a total possible range of 0-40. Higher scores indicate greater burnout, indicating lower well-being

SECONDARY OUTCOMES:
Change in time spent on documentation outside work hours | Baseline to 24 weeks
  Providers will track amount of time spent on EHR (electronic health records) outside of scheduled patient hours per 8 hours of patient scheduled time
Change in task load | Baseline to 24 weeks
  Hours spent on documentation per 8 hours of scheduled patient time
Change in meaningfulness of work | Baseline to 24 weeks
  Meaningfulness of work is a 4-item questionnaire, where each question is scored on a 0-4 Likert scale. Total possible scores range from 0-16, with higher scores indicating lower sense of meaningfulness of work.
Change in meaningful relationships | Baseline to 24 weeks
  Using the Professional Well-Being Academic Consortium Survey Measures, the negative impact of work on relationships index is a 4-item questionnaire. Each question is scored on a 0-4 Likert scale, with total possible scores ranging from 0-16. Higher scores indicate less meaningful relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Majid Afshar, MD, MS, Principal Investigator — University of Wisconsin, Madison; Joel Gordon, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of the UW Learning Health System, the data queries, data dictionary, and data procedure will be mirrored over from the UW Health GitHub instance to SMPH GitLab instance for secondary research use. All patient data except timestamps will be deidentified (limited dataset) and managed and stored on SMPH servers and devices and provided through Clinical Research Data Service (CRDS) team in ICTR's Center for Health Informatics Institute and the UW SMPH Honest Broker. Provider data will be stored with identifiers for the follow-up focus groups and interviews.
Supporting Information: Study Protocol
Time Frame: Duration of storage will be at least 10 years.
Access Criteria: Access to data and recordings and security measures will require IRB approval and request through CRDS.
URL: https://ictr.wisc.edu/consults/biomedical-informatics/

REFERENCES:
- [Derived] Afshar M, Baumann MR, Resnik F, Hintzke J, Sullivan AG, Wills G, Lemmon K, Dambach J, Ann Mrotek L, Quinn M, Abramson K, Kleinschmidt P, Brazelton TB, Leaf MA, Twedt H, Kunstman D, Patterson B, Liao F, Rasmussen S, Burnside ES, Goswami C, Gordon J. A Pragmatic Randomized Controlled Trial of Ambient Artificial Intelligence to Improve Health Practitioner Well-Being. NEJM AI. 2025 Dec;2(12):10.1056/aioa2500945. doi: 10.1056/aioa2500945. Epub 2025 Nov 26. PMID 41625485
- [Derived] Afshar M, Resnik F, Baumann MR, Hintzke J, Lemmon K, Sullivan AG, Shah T, Stordalen A, Oberst M, Dambach J, Mrotek LA, Quinn M, Abramson K, Kleinschmidt P, Brazelton T, Twedt H, Kunstman D, Wills G, Long J, Patterson BW, Liao FJ, Rasmussen S, Burnside E, Goswami C, Gordon JE. A Novel Playbook for Pragmatic Trial Operations to Monitor and Evaluate Ambient Artificial Intelligence in Clinical Practice. NEJM AI. 2025 Sep;2(9):10.1056/aidbp2401267. doi: 10.1056/aidbp2401267. Epub 2025 Aug 28. PMID 40959192
- [Derived] Afshar M, Resnik F, Baumann MR, Hintzke J, Lemmon K, Sullivan AG, Shah T, Stordalen A, Oberst M, Dambach J, Mrotek LA, Quinn M, Abramson K, Kleinschmidt P, Brazelton T, Twedt H, Kunstman D, Wills G, Long J, Patterson BW, Liao FJ, Rasmussen S, Burnside E, Goswami C, Gordon JE. A Novel Playbook for Pragmatic Trial Operations to Monitor and Evaluate Ambient Artificial Intelligence in Clinical Practice. medRxiv [Preprint]. 2025 Aug 14:2024.12.27.24319685. doi: 10.1101/2024.12.27.24319685. PMID 39763559